CLINICAL TRIAL: NCT05259826
Title: Improving the Diagnosis of Food Allergy and Food Intolerance by Determining Mucosal IgE and Inflammatory Markers and Validating With Intestinal in Vitro Organoids
Brief Title: Mucosal IgE to Improve Diagnosis of Food Allergy and Food Hypersensitivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, yurdagül zopf, Professor Dr., University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-474-B
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Food Allergy; Food Hypersensitivity
Keywords: mucosal IgE; inflammation parameter
MeSH Terms: conditions — Food Hypersensitivity | interventions — Chorionic Villi Sampling

STUDY DESIGN:
Intervention Model Description: Data derived from patients with food hypersensitivity will be compared with data of healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with food hypersensitivity (Experimental)
  Interventions: Other: biopsy sampling
- healthy controls (Experimental)
  Interventions: Other: biopsy sampling

INTERVENTIONS:
Other: biopsy sampling — 1. Biopsies are homogenised in buffer and used for the determination of mucosal IgE and inflammatory parameters.
  2. Biopsies are used to isolate organoids, stimulate them with blood cells and food antigens and to study gene and protein expression.

SUMMARY:
Aim of the study is to improve the diagnosis of food allergy and hypersensitivity. Intestinal homogenates will be used to determine total IgE, specific IgE, tryptase, histamine and inflammation parameters (IFNgamma, TNFalpha). These data will be correlated with serum values and disease status. In addition, organoids from duodenal tissue will be isolated and cultured in vitro and stimulated with the major food allergens. The gene and protein expression will be checked to identify relevant biomarkers.

DETAILED DESCRIPTION:
Food intolerances (FI) show an increasing prevalence and represent a particular challenge in clinical practice. The symptoms of a predominantly gastrointestinally mediated food allergy (FA) are similar to the symptoms of other FI (e.g. carbohydrate malabsorption, gluten sensitivity, histamine intolerance, irritable bowel syndrome), so that diagnosis is difficult and often delayed.

Well-evaluated methods for the clarification of an allergic disease are serological screening (IgE against food products or other cross-reacting allergens) and skin prick tests. However, these methodes have their limitations in the diagnosis of seronegative or mainly gastrointestinal-mediated FI. Patients often associate the consumption of certain foods with the clinical symptoms, which often leads to strict self-imposed elimination diets, but rarely to the correct identification of the triggering food.

In a pilot study, the investigators showed that patients with gastrointestinal FI have elevated mucosal IgE levels and TNF using homogenates from intestinal biopsies. Another patient subgroup could be identified that showed low allergic parameters (low mucosal IgE, low TNF) but high mucosal interferon levels, indicating a non-specific inflammation.

In this study, mucosal IgE, tryptase, histamine, IL4, and inflammatory parameters (e.g. TNF, IFN) from different areas of the gastrointestinal tract will be determined in a larger collective. Furthermore, organoids are cultured in vitro from duodenal tissue samples, incubated with blood cells and stimulated with food allergens. The titres of specific IgE from the mucosal homogenates will be correlated with serum levels and organoid stimulation results to identify relevant biomarkers. Microbiome and metabolome analyses will provide information about the intestinal flora in FI.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* patients with suspected food allergy or hypersensitivity
* healthy controls with indications for endoscopic diagnostics, e.g. tumour history within the family, exclusion of gastritis

Exclusion Criteria:

* pregnant person

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Determination of mucosal IgE to identify patients with gastrointestinal food allergy | 3 years
  Homogenates of mucosal biopsies will be checked for IgE levels

SECONDARY OUTCOMES:
Identification of patients with food hypersensitivity | 3 years
  Homogenates of mucosal biopsies will be checked for inflammatory parameters (TNF, IFN)
Correlation of mucosal IgE and inflammatory parameters with data from organoids | 3 years
  Organoids are isolated from intestinal biopsies, co-cultured with blood cells and stimulated with food antigens. Gene and protein expression will be correlated with mucosal IgE and inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine 1, Hector Center for Nutrition, Exercise and Sports, Friedrich-Alexander-University Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No